CLINICAL TRIAL: NCT04818671
Title: A Long-Term, Single-Arm, Open-label, Multicenter Phase 3 Study to Evaluate the Safety and Tolerability of Multiple Subcutaneous Injections of Efgartigimod PH20 SC in Patients With Generalized Myasthenia Gravis
Brief Title: Evaluating the Long-Term Safety and Tolerability of Efgartigimod PH20 SC Administered Subcutaneously in Patients With Generalized Myasthenia Gravis
Acronym: ADAPTSC+
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: argenx (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARGX-113-2002
Record Dates: First submitted 2021-03-11; First posted 2021-03-26 (Actual); Results first posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Generalized Myasthenia Gravis
MeSH Terms: conditions — Myasthenia Gravis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- efgartigimod PH20 SC (Experimental): Patients receiving efgartigimod PH20 subcutaneous (SC) treatment
  Interventions: Biological: efgartigimod PH20 SC

INTERVENTIONS:
Biological: efgartigimod PH20 SC — Subcutaneous injection with efgartigimod PH20 SC

SUMMARY:
The purpose of this study is to evaluate the long-term safety and tolerability of efgartigimod PH20 SC 1000 mg, and the clinical efficacy, PD, pharmacokinetics (PK), immunogenicity, impact on the quality of life (QoL) of the participants, treatment satisfaction, and administration method preference, and the feasibility of self- and caregiver-supported administration of the SC injection.

Treatment duration: 3-week treatment periods, repeated as needed with at least 28 days in between treatment periods

Health measurements: total levels of immunoglobulin G (IgG), Acetylcholine receptor binding autoantibodies (AChR-Ab) levels, Myasthenia Gravis Activities of Daly Living (MG-ADL).

ELIGIBILITY:
Inclusion Criteria:

1. Must be capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.
2. Previously participated in antecedent studies ARGX-113-2001 or ARGX-113-1705 and are eligible for roll over.
3. Contraceptive use by men and women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies and:

   * Women of Child bearing potential (WOCBP) must have a negative urine pregnancy test at baseline before investigational medicinal product (IMP) can be administered.

Exclusion Criteria:

1. The participant was discontinued early from studies ARGX-113-2001 or ARGX-113-1705, unless the reason for discontinuation from study ARGX-113-1705 was to roll over into study ARGX-113-2002.

   a. Participants who, in the investigator's judgment, are not benefiting from efgartigimod IV in study ARGX-113-1705 Part B are not eligible for roll over into ARGX-113-2002.
2. Are pregnant or lactating, or intend to become pregnant during the study or within 90 days after the last dose of investigational medicinal product (IMP)
3. Has any of the following medical conditions:

   1. Clinically significant uncontrolled chronic bacterial, viral, or fungal infection at roll-over
   2. Any other known autoimmune disease that, in the opinion of the investigator, would interfere with accurate assessment of clinical symptoms of myasthenia gravis or put the participant at undue risk
   3. History of malignancy unless deemed cured by adequate treatment with no evidence of reoccurrence for ≥3 years before the first administration of investigational medicinal product (IMP).

      Participants with the following cancers can be included at any time:
      * adequately treated basal cell or squamous cell skin cancer
      * carcinoma in situ of the cervix
      * carcinoma in situ of the breast
      * incidental histological findings of prostate cancer (TNM classification of malignant tumors stage T1a or T1b)
   4. Clinical evidence of other significant serious diseases, or the participant has had a recent major surgery, or who have any other condition that, in the opinion of the investigator, could confound the results of the study or put the participant at undue risk
4. Received a live-attenuated vaccine within 28 days prior to study entry or plan to receive a live-attenuated vaccine during the study
5. A known hypersensitivity reaction to efgartigimod, rHuPH20, or any of its excipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2021-04-26 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (47):
- United States (13):
  - Investigator site 6 - US0010032, Carlsbad, California
  - Investigator Site 47 - US0010021, Palo Alto, California
  - Investigator Site 45 - US0010108, Boca Raton, Florida
  - Investigator site 4 - US0010110, Port Charlotte, Florida
  - Investigator Site 39 - US0010006, Tampa, Florida
  - Investigator Site 41 - US0010015, Kansas City, Kansas
  - Investigator Site 46 - US0010111, Amherst, New York
  - Investigator Site 38 - US0010003, Chapel Hill, North Carolina
  - Investigator Site 44 - US0010077, Durham, North Carolina
  - Investigator Site 42 - US0010019, Cleveland, Ohio
  - Investigator site 7 - US0010008, Cordova, Tennessee
  - Investigator Site 43 - US0010066, Austin, Texas
  - Investigator Site 40 - US0010009, San Antonio, Texas
- Investigator site 5 - BE0320007, Ghent, Belgium
- Investigator site 24 - CZ4200005, Brno, Czechia
- Georgia (5):
  - Investigator Site 32 - GEO9950004, Tbilisi, K'alak'i T'bilisi
  - Investigator Site 33 - GEO9950016, Tbilisi, K'alak'i T'bilisi
  - Investigator site 2 - GEO9950002, Tbilisi
  - Investigator Site 1 - GEO9950001, Tbilisi
  - Investigator site 3 - GEO9950003, Tbilisi
- Germany (2):
  - Investigator Site 25 - DE490006, Berlin
  - Investigator Site 26 - DE490009, Münster
- Hungary (2):
  - Investigator site 10 - HU0360013, Budapest
  - Investigator site 9 - HU0360012, Budapest
- Italy (3):
  - Investigator site 11 - IT0390003, Milan
  - Investigator Site 34 - IT0390007, Napoli
  - Investigator Site 35 - IT0390008, Roma
- Japan (8):
  - Investigator site 12 - JP0810002, Chiba, Chiba-Shi
  - Investigator Site 36 - JP0810055, Sapporo, Hokkaido
  - Investigator site 8 - JP0810004, Hanamaki, Iwate
  - Investigator Site 28- JP0810059, Ōta-ku, Tokyo
  - Investigator site 14 - JP0810007, Osaka
  - Investigator Site 27 - JP0810008, Sapporo
  - Investigator site 13 - JP0810005, Sendai
  - Investigator site 15 - JP0810009, Tokyo
- Investigator site 16 - NL0310001, Leiden, Netherlands
- Poland (6):
  - Investigator site 17 - PL0480001, Gdansk
  - Investigator site 19 - PL0480007, Katowice
  - Investigator site 22 - PL0480065, Krakow
  - Investigator site 18 - PL0480005, Krakow
  - Investigator site 20 - PL0480018, Lublin
  - Investigator site 21 - PL0480022, Warsaw
- Russia (2):
  - Investigator Site 29- RU0070002, Novosibirsk
  - Investigator Site 30 - RU0070014, Saint Petersburg
- Spain (3):
  - Investigator Site 37 - ES0340021, Barcelona
  - Investigator Site 31 - ES0340038, Barcelona
  - Investigator site 23 - ES0340039, Valencia

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 47 sites that enrolled participants in 12 countries. A total of 184 participants rolled over from ARGX-113-2001 and ARGX-113-1705, of whom 180 participants were exposed to efgartigimod PH20 SC treatment.
Pre-assignment Details: All participants were adults with gMG who participated in ARGX-113-2001 or ARGX-113-1705. No randomization or blinding was performed because this was an open-label study.
Groups:
- Efgartigimod PH20 SC: Patients receiving efgartigimod PH20 subcutaneous (SC) treatment; efgartigimod PH20 SC: efgartigimod for SC administration coformulated with recombinant human hyaluronidase PH20
Period: Overall Study
Arm/Group | Efgartigimod PH20 SC
Started | 180
Completed | 138
Not Completed | 42
Not completed — Withdrawal by Subject | 16
Not completed — Adverse Event | 5
Not completed — Lack of Efficacy | 5
Not completed — Death | 4
Not completed — Physician Decision | 4
Not completed — Requires Prohibited Medication | 4
Not completed — Lost to Follow-up | 2
Not completed — Approved Drug Available for Indication | 1
Not completed — Sponsor Request | 1

BASELINE CHARACTERISTICS:
Arm/Group | Efgartigimod PH20 SC
Number analyzed (Participants) | 180
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 139
  >=65 years | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.8 (15.50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 119
  Male | 61
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 16
  Black or African American | 2
  White | 161
  Multiple | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 8
  Not Hispanic or Latino | 172

OUTCOME MEASURES:

1. Primary Outcome: Number of AEs, SAEs and AESIs
Description: Adverse events, Serious Adverse event and Adverse events of special interest. Adverse events in the 'Infections and infestations' SOC were defined as AESIs because efgartigimod causes a transient reduction in total IgG levels.
Time Frame: Up to 3.5 years
Population: Safety analysis set: all participants who were exposed to efgartigimod PH20 SC in this study
Measure: Number; unit: events
Arm/Group | Efgartigimod PH20 SC
Number analyzed (Participants) | 180
events
  Number of AEs | 3325
  Number of SAEs | 107
  Number of AESIs | 420

2. Secondary Outcome: MG-ADL Total Score Changes From Baseline
Description: The Myasthenia Gravis Activities of Daily Living (MG-ADL) is an 8-item patient-reported scale that assesses MG symptoms and their effects on daily activities. It evaluates a participant's capacity to perform different activities in their daily life. The total score ranges from 0 to 24 with higher scores indicating more impairment.
Time Frame: Up to week 4 of the first cycle
Population: Safety analysis set: all participants who were exposed to efgartigimod PH20 SC in this study. Only participants with an assessment at baseline and the respective weeks of first cycle are reported in each row.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Efgartigimod PH20 SC
Number analyzed (Participants) | 180
score on a scale
  Cycle 1, Week 1 | -2.2 (0.20)
  Cycle 1, Week 2: number analyzed (Participants) | 176
  Cycle 1, Week 2 | -3.4 (0.21)
  Cycle 1, Week 3: number analyzed (Participants) | 176
  Cycle 1, Week 3 | -3.9 (0.22)
  Cycle 1, Week 4: number analyzed (Participants) | 170
  Cycle 1, Week 4 | -4.0 (0.23)

3. Secondary Outcome: Percent Change in Total IgG Levels From Baseline
Description: IgG: immunoglobulin G
Time Frame: Up to week 4 of the first cycle
Population: Safety analysis set: all participants who were exposed to efgartigimod PH20 SC in this study. Only participants with an assessment at baseline and week 4 of the first cycle are reported.
Measure: Mean (Standard Error); unit: Percent change
Arm/Group | Efgartigimod PH20 SC
Number analyzed (Participants) | 164
Percent change | -62.6 (0.93)

4. Secondary Outcome: Percent Change in AChR-Ab From Baseline in AChR-Ab Seropositive Participants
Description: AchR-Ab: anti-acetylcholine receptor antibodies.
Time Frame: Up to week 4 of the first cycle
Population: as for outcome 3
Measure: Mean (Standard Error); unit: Percent change
Arm/Group | Efgartigimod PH20 SC
Number analyzed (Participants) | 124
Percent change | -57.6 (2.29)

5. Secondary Outcome: Efgartigimod Serum Concentrations
Time Frame: Up to week 4 of the first cycle
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Efgartigimod PH20 SC
Number analyzed (Participants) | 141
ng/mL | 21693 (8242)

6. Secondary Outcome: Incidence of ADAs Against Efgartigimod Over Time
Description: ADA: Anti-drug antibodies.
Time Frame: Up to 3.5 years
Population: Safety analysis set: all participants who were exposed to efgartigimod PH20 SC in this study. The number analyzed is the total number of ADA evaluable participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Efgartigimod PH20 SC
Number analyzed (Participants) | 178
Participants | 35

7. Secondary Outcome: Incidence of NAbs Against Efgartigimod Over Time
Description: NAbs: neutralizing antibodies
Time Frame: Up to 3.5 years
Population: Safety analysis set: all participants who were exposed to efgartigimod PH20 SC in this study. The number analyzed is the total number of NAb-evaluable participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Efgartigimod PH20 SC
Number analyzed (Participants) | 178
Participants | 11

8. Secondary Outcome: Incidence of Antibodies Against rHuPH20 Over Time
Time Frame: Up to 3.5 years
Population: Safety analysis set: all participants who were exposed to efgartigimod PH20 SC in this study. The number analyzed is the total number of rHuPH20 Ab evaluable participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Efgartigimod PH20 SC
Number analyzed (Participants) | 170
Participants | 49

9. Secondary Outcome: Incidence of NAbs Against rHuPH20 Over Time
Description: NAbs: neutralizing antibodies
Time Frame: Up to 3.5 years
Population: Safety analysis set: all participants who were exposed to efgartigimod PH20 SC in this study. The number analyzed is the total number of rHuPH20 NAb-evaluable participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Efgartigimod PH20 SC
Number analyzed (Participants) | 167
Participants | 1

10. Secondary Outcome: Changes in Total MG-QoL15r From Baseline
Description: Myasthenia Gravis Quality of Life 15 item scale revised (MG-QoL 15r) scores range from 0 to 30 with a higher score representing more severe symptoms.
Time Frame: Up to week 4 of the first cycle
Population: as for outcome 2
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Efgartigimod PH20 SC
Number analyzed (Participants) | 180
score on a scale
  Cycle 1, Week 1: number analyzed (Participants) | 179
  Cycle 1, Week 1 | -2.5 (0.29)
  Cycle 1, Week 2: number analyzed (Participants) | 175
  Cycle 1, Week 2 | -3.7 (0.34)
  Cycle 1, Week 3: number analyzed (Participants) | 175
  Cycle 1, Week 3 | -4.5 (0.38)
  Cycle 1, Week 4: number analyzed (Participants) | 168
  Cycle 1, Week 4 | -4.7 (0.39)

11. Secondary Outcome: Changes in EQ-5D-5L VAS Score From Baseline
Description: EuroQoL 5 Dimensions 5-Level (EQ-5D-5L) visual analog scale (VAS) scores range from 0 to 100 with a higher score representing better health.
Time Frame: Up to week 4 of the first cycle
Population: as for outcome 3
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Efgartigimod PH20 SC
Number analyzed (Participants) | 169
score on a scale | 13.9 (1.32)

12. Secondary Outcome: Percent of Participants or Caregivers by Number of Training Visits Needed to be Competent to Start Self- or Caregiver-Supported Administration
Time Frame: Up to 3.5 years
Population: Safety analysis set: all participants who were exposed to efgartigimod PH20 SC in this study. The number analyzed is the total number of participants adequately trained and capable of doing self- or caregiver-supported administrations.
Measure: Number; unit: Percent of participants
Arm/Group | Efgartigimod PH20 SC
Number analyzed (Participants) | 166
Percent of participants
  0 visits | 4.8
  1 visit | 45.8
  2 visits | 13.9
  3 visits | 11.4
  4 visits | 12.7
  5 visits | 1.8
  6 visits | 5.4
  9 visits | 1.2
  11 visits | 0.6
  12 visits | 0.6
  22 visits | 0.6
  37 visits | 0.6
  42 visits | 0.6

13. Secondary Outcome: Percent of Self- or Caregiver-supported Study Drug Administration Among All Study Treatment Visits at Home
Time Frame: Up to 3.5 years
Population: Safety analysis set: all participants who were exposed to efgartigimod PH20 SC in this study.
Measure: Number; unit: Percent
Arm/Group | Efgartigimod PH20 SC
Number analyzed (Participants) | 180
Percent | 49.2

ADVERSE EVENTS:
Time Frame: 3.5 years
Description: Any clinically significant changes occurring during the study were reported as adverse events.
Arm/Group | Efgartigimod PH20 SC
All-Cause Mortality (participants affected / at risk) | 5/180
Serious Adverse Events (participants affected / at risk) | 55/180
Other Adverse Events (participants affected / at risk) | 167/180
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Efgartigimod PH20 SC (N=180)
Anaemia (Blood and lymphatic system disorders) | 1
Acute myocardial infarction (Cardiac disorders) | 1
Angina unstable (Cardiac disorders) | 2
Cardiac arrest (Cardiac disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 2
Diplopia (Eye disorders) | 1
Retinal detachment (Eye disorders) | 1
Vitreous haemorrhage (Eye disorders) | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Inguinal hernia (Gastrointestinal disorders) | 1
Intestinal perforation (Gastrointestinal disorders) | 1
Terminal ileitis (Gastrointestinal disorders) | 1
Anal abscess (Infections and infestations) | 1
Bacteraemia (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 2
Cellulitis gangrenous (Infections and infestations) | 1
COVID-19 (Infections and infestations) | 4
COVID-19 pneumonia (Infections and infestations) | 1
Diarrhoea infectious (Infections and infestations) | 1
Diverticulitis (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Orchitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 7
Rotavirus infection (Infections and infestations) | 1
Sepsis (Infections and infestations) | 2
Urinary tract infection (Infections and infestations) | 1
Viral infection (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 1
Post procedural complication (Injury, poisoning and procedural complications) | 1
Rib fracture (Injury, poisoning and procedural complications) | 2
Shunt occlusion (Injury, poisoning and procedural complications) | 1
Shunt stenosis (Injury, poisoning and procedural complications) | 1
Spinal fracture (Injury, poisoning and procedural complications) | 1
Tendon injury (Injury, poisoning and procedural complications) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Enthesopathy (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Spondyloarthropathy (Musculoskeletal and connective tissue disorders) | 1
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Rectal cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Renal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Thymoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Coma (Nervous system disorders) | 1
Myasthenia gravis (Nervous system disorders) | 11
Myasthenia gravis crisis (Nervous system disorders) | 4
Syncope (Nervous system disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4
Umbilical hernia repair (Surgical and medical procedures) | 1
Uterine polypectomy (Surgical and medical procedures) | 1
Brachiocephalic vein stenosis (Vascular disorders) | 1
Hypertension (Vascular disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Efgartigimod PH20 SC (N=180)
Anaemia (Blood and lymphatic system disorders) | 18
Iron deficiency anaemia (Blood and lymphatic system disorders) | 13
Cataract (Eye disorders) | 9
Abdominal pain upper (Gastrointestinal disorders) | 11
Diarrhoea (Gastrointestinal disorders) | 32
Nausea (Gastrointestinal disorders) | 16
Fatigue (General disorders) | 10
Influenza like illness (General disorders) | 14
Injection site bruising (General disorders) | 24
Injection site erythema (General disorders) | 55
Injection site haematoma (General disorders) | 10
Injection site pain (General disorders) | 22
Injection site pruritus (General disorders) | 21
Injection site rash (General disorders) | 15
Injection site reaction (General disorders) | 10
Injection site swelling (General disorders) | 11
Pyrexia (General disorders) | 9
Bronchitis (Infections and infestations) | 9
COVID-19 (Infections and infestations) | 52
Influenza (Infections and infestations) | 9
Nasopharyngitis (Infections and infestations) | 36
Upper respiratory tract infection (Infections and infestations) | 32
Urinary tract infection (Infections and infestations) | 16
Contusion (Injury, poisoning and procedural complications) | 9
Activated partial thromboplastin time prolonged (Investigations) | 12
Arthralgia (Musculoskeletal and connective tissue disorders) | 17
Back pain (Musculoskeletal and connective tissue disorders) | 22
Muscle spasms (Musculoskeletal and connective tissue disorders) | 11
Pain in extremity (Musculoskeletal and connective tissue disorders) | 11
Dizziness (Nervous system disorders) | 13
Headache (Nervous system disorders) | 48
Myasthenia gravis (Nervous system disorders) | 18
Cough (Respiratory, thoracic and mediastinal disorders) | 12
Hypertension (Vascular disorders) | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-02-02): https://cdn.clinicaltrials.gov/large-docs/71/NCT04818671/Prot_000.pdf
  • Statistical Analysis Plan (2025-01-31): https://cdn.clinicaltrials.gov/large-docs/71/NCT04818671/SAP_001.pdf